CLINICAL TRIAL: NCT00993135
Title: Renal Dysfunction With Low to Intermediate Dose Methotrexate in Acute Lymphoblastic Leukemia Treatment
Brief Title: Kidney Dysfunction in Children and Young Adults Who Have Received Methotrexate for Acute Lymphoblastic Leukemia
Status: Completed | Type: Observational
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000652517; P30CA068485 (NIH); VU-VICC-PED-0913; IRB# 081330
Record Dates: First submitted 2009-10-09; First posted 2009-10-12 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Leukemia; Renal Toxicity
Keywords: renal toxicity; childhood acute lymphoblastic leukemia; adult acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Methotrexate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: methotrexate
Other: medical chart review
Procedure: assessment of therapy complications

SUMMARY:
RATIONALE: Gathering information about how often kidney dysfunction occurs in children and young adults receiving methotrexate for acute lymphoblastic leukemia may help doctors learn more about the disease and plan the best treatment.

PURPOSE: This research study is looking at kidney dysfunction in children and young adults who have received low-dose or intermediate-dose methotrexate for acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Examine the incidence of renal dysfunction in children and young adults being treated for acute lymphoblastic leukemia with low- to intermediate-dose methotrexate.

OUTLINE: Medical charts are reviewed to obtain the following information: gender, age, diagnosis, regimen, day of therapy, renal function, creatinine level, mucositis, skin sloughing, methotrexate level at highest level, and number of days after intravenous methotrexate.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of acute lymphoblastic leukemia

  * Receiving low- to intermediate-dose methotrexate or received treatment (chemotherapy and/or radiation) at Vanderbilt Children's Hospital

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2008-12; Primary Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Incidence of renal dysfunction in children and young adults being treated for acute lymphoblastic leukemia with low- to intermediate-dose methotrexate

CONTACTS AND LOCATIONS:
Overall Officials: Pinki Prasad, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (2):
- United States (2):
  - Vanderbilt-Ingram Cancer Center - Cool Springs, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee